CLINICAL TRIAL: NCT01624623
Title: Post-prostatectomy Daily Target Guided Radiotherapy Using Real-Time, State-of-the-Art Motion Tracking With the Calypso 4D Localization System: A Feasibility Study
Brief Title: Daily Target Guided Radiation Therapy Using the Calypso 4D Localization System in Patients Who Have Had a Prostatectomy for Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dusten Macdonald, MD, MD, MC, Madigan Army Medical Center
Other Study IDs: W81XWH-08-2-0174, A-15214.3; 210016 (Other: Madigan Army IRB)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Prostate Cancer
Keywords: radiation; Calypso; prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will evaluate the daily use of a unique daily organ tracking system on target localization in patients treated with radiation therapy after radical prostatectomy for prostate cancer.

Improved coverage of the target volume with radiotherapy could result in improved cancer control rates and decreased coverage of surrounding structures potentially decreasing treatment toxicity.

DETAILED DESCRIPTION:
This prospective study evaluates the clinical utility of a novel real-time localization system of the prostate bed during adjuvant or salvage radiotherapy after radical prostatectomy. This study will also determine positioning errors using daily cone-beam computed tomography in patients set up with the Calypso 4D Localization System. Subjects will have Beacon® Transponders implanted into the prostate bed. The Calypso 4D Localization System will localize the position of the prostate bed. Cone beam CT will be used daily to measure inter-transponder distance. The Calypso system will also track the prostate bed position in real time during the entire radiation treatment. The treatments will be adjusted as required to ensure accurate treatment of the clinical target volume. The time of, the number, and extent of adjustments will be recorded for analysis.

Daily cone-beam computed tomography images will also be retrospectively analyzed to assess for adequate target coverage. The analysis will be performed retrospectively through manual 3-D registration of the cone-beam CT dataset with the treatment planning CT scan. This information will determine the margins necessary for the PTV using the Calypso 4D Localization System and potentially may allow a reduction in the PTV volumes on future studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate initially managed with prostatectomy with a detectable PSA, positive surgical margins, or extra-prostatic extension.
* Ability to comply with study schedule
* Age 40 or older
* Zubrod PS 0 or 1 (appendix 1)
* Signed informed consent

Exclusion Criteria:

* Node positive or metastatic prostate cancer
* History of prior pelvic radiotherapy
* History of abdominoperineal resection
* History of inflammatory bowel disease or connective tissue disease
* History of bleeding disorder or any active anticoagulant or anti-platelet medication which cannot be discontinued safely for transponder placement.
* PT or INR outside normal range for institution
* Active implanted devices such as cardiac pacemakers and automatic defibrillators.
* Prosthetic implants in the pelvic region that contain metal or conductive materials (eg., an artificial hip).
* Patients with maximum anterior-posterior separation through the torso minus the height of the center of the prostate greater than 17 cm (technical reason for Calypso System, see appendix 5).
* History of HIV infection

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include high risk patients referred for adjuvant or salvage radiation therapy after radical prostatectomy based upon the presence of unfavorable characteristics after prostatectomy, which include positive surgical margins, extracapsular extension of disease, or immediately detectable PSA.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Interfraction prostate bed motion | Approximately 7.5 weeks (36-39 fractions per pt.)
  For each fraction, measurements from the registered CTV (clinical target volume) at the midline will be obtained to structures at 3 points to assess for the degree of motion.
  1. Inferior (defined as 8 mm below VUA)
  2. Superior (top of seminal vesicle remnant or superior most CTV slice)
  3. Middle (defined as the slice equally distant from the inferior and superior slices above)
Intrafraction prostate bed motion | Approximately 7.5 weeks (36-39 fractions per pt.)
  Calypso session reports measuring intrafraction motion in x,y,z axis will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Dusten Macdonald, MD, Principal Investigator — Department of the Army
Locations (1):
- Madigan Healthcare System, Tacoma, Washington, United States